CLINICAL TRIAL: NCT03767049
Title: Readmissions of Lung Transplant Patients in the Intensive Care Unit
Brief Title: Readmissions of Lung Transplant Patients in ICU.
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Other Study IDs: PR(AG)101/2012
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Lung Transplant; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung transplant patients readmitted in ICU
  Interventions: Other: Colection of clinical data

INTERVENTIONS:
Other: Colection of clinical data — Colection of clinical data

SUMMARY:
A multi-centre, prospective and observational study was carried out from August 2012 to June 2016 in five Spanish tertiary-care university hospitals with well-established lung transplant programs: Vall d'Hebron (Barcelona), Marqués de Valdecilla (Santander), 12 de Octubre (Madrid), CHUAC (A Coruña), and Reina Sofía (Córdoba).

The study population comprised all consecutive adult lung transplant recipients who required ICUr (after >7 days post-transplant discharge from ICU) during august 2012 - June 2016 (4-yr period).

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult lung transplant recipients who required ICU readmission (after >7 days post-transplant discharge from ICU) during august 2012 - June 2016 (4-yr period).

Exclusion Criteria:

* ICU readmission < 8 days post-transplant discharge from ICU.
* ICU readmission for early postoperative care following lung transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant recipients who required ICU readmission.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Causes of ICU readmission in LT adults | Augist 1. 2012 - June 30, 2016
  To assess the principal causes of ICU readmission in LT adults.
Predictors of ICU and hospital mortality. | Augist 1. 2012 - June 30, 2016
  To identify potential predictors of ICU and hospital mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Cristopher Alan Mazo Torre, MD, Study Chair — 0

IPD SHARING:
Plan to Share IPD: Undecided